CLINICAL TRIAL: NCT01617811
Title: Effects of Epidural Anesthesia and Analgesia on Postoperative Metabolic, Immune Function and Hemodynamic Changes of Open Liver Resection
Brief Title: Effect of Epidural Anesthesia and Analgesia on Patients' Outcomes After Liver Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Chun-Yan Yan, M.D. , Ph.D, Sir Run Run Shaw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20120530; No. 2009R50040 (Other Grant/Funding Number: Foundation of Science and Technology Department of Zhejiang)
Record Dates: First submitted 2012-06-05; First posted 2012-06-12 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Hepatectomy
MeSH Terms: interventions — Anesthesia, Epidural; Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: epidural anesthesia and analgesia — A thoracic epidural catheter (T8-10) was placed in group E. A bolus of 8ml 1% lidocaine with 0.375% ropivacaine was administered 15min before skin incision, followed by 5-8 ml/hr infusion during surgery in group E.
  Postoperative analgesia by PCEA in group E (concentration: 0.1% ropivacaine + 0.1μg/ml sufentanil, loading dose: 4ml, infusion rate: 8ml/hr, bolus: 4ml, 1hr limit: 16ml) and lasting for 48hr and PCIA in group G (concentration: 1μg/ml sufentanil, loading dose: 4ml, bolus: 2ml, 4hr limit: 30ml).
  Both group received general anesthesia maintaining with 1-2% end tidal sevoflurane together with TCI of propofol (target plasma concentration, 2-3µg/ml), continuous infusion of remifentanil (0.10 - 0.20 μg/kg/min) and cis-atracurium intermittently as needed.

SUMMARY:
The purpose of this study is to analyze the effects of epidural anesthesia and analgesia on intraoperative clinical outcome, postoperative recovery, metabolic changes, and immune functions of the patients receiving open liver resection.

ELIGIBILITY:
Inclusion Criteria:

* left hemihepatectomy left lateral sectionectomy clinical diagnosis of hepatolithiasis

Exclusion Criteria:

* abnormal coagulation tests diabetes mellitus significant cirrhosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes during and after open liver resection | participants will be followed for the duration of hospital stay, an expected average of 4 weeks
  intraoperative outcome including operation time, liver resection time, estimated blood loss, urine output, etc during operation. PACU recovery, pain score, liver and gastrointestinal function, hospital stay time,etc assessed.
  Before operation, right after operation(0), and 3hr, 12hr, 24hr, 72hrs after operation, blood glucose and insulin was measured.

SECONDARY OUTCOMES:
Cytokine change in perioperation of open liver resection | Before operation, within 5 days after operation
  Before operation and 0, 3hr, 12hr, 24hr, D3, D5 after operation, serum IL-1β, IFN-γ, IL-4, IL-10 and TGF-β by microassay.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China